CLINICAL TRIAL: NCT06366698
Title: Randomized Control Trial: Intravenous Iron Versus Oral Iron for the Treatment of Iron Deficiency Anemia in Pregnancy
Brief Title: Intravenous Iron Versus Oral Iron for the Treatment of Iron Deficiency Anemia
Acronym: IDA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-55
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Iron Deficiency Anemia of Pregnancy
Keywords: Anemia; Iron deficiency; Pregnancy; Intravenous iron
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — Ferric Oxide, Saccharated; Injections; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Patients are initially randomized to either PO or IV iron, after the initial 4-week treatment patients in the PO iron group can switch to IV iron if labs continue to show persist iron deficiency anemia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous iron (Active Comparator): Venofer 200 mg will be given every other day until the patient reaches their calculated in deficit dose. The does of IV iron will be calculated according to the Ganzoni formula: total iron dose (mg) = body weight (kg) x (target Hgb - baseline Hgb (g/dL)) × 0.24 + 500 mg.14 Our target Hgb will be 11.0 g/dL. The determination of the treatment duration and dosage will be based on the calculation of the iron deficit.
  Interventions: Drug: Venofer 200 MG Per 10 ML Injection
- Oral iron (Placebo Comparator): Ferrous sulfate 325 mg orally every other day on an empty stomach with lemon/orange water until delivery.
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Venofer 200 MG Per 10 ML Injection — 200 mg IV every 2 days until the targeted dose
  Other Names: Iron sucrose
  Arms: Intravenous iron
Drug: Ferrous sulfate — Take 1 tablet every other day with lemon/orange juice
  Arms: Oral iron

SUMMARY:
This study aims to assess whether administering intravenous iron early in pregnancy, compared to standard oral iron treatment, can enhance hemoglobin levels before delivery and reduce the need for blood transfusions in patients with iron deficiency anemia. Patients diagnosed with iron deficiency anemia were randomly assigned to receive either oral or intravenous iron. Before treatment initiation, patients completed a symptom questionnaire baseline hemoglobin, and ferritin levels were measured. Follow-up visits occurred four weeks later and at 24 to 28 weeks gestation, involving reassessment of symptoms, laboratory testing, and monitoring of treatment adherence. Final hemoglobin levels were determined before delivery, and data on the need for blood transfusion at delivery were recorded.

DETAILED DESCRIPTION:
Iron deficiency anemia is a prevalent health concern affecting approximately a quarter of the global population. In specific high-risk subgroups such as pregnancy, the occurrence of anemia is even higher. This condition is associated with adverse outcomes such as increased risks of blood transfusion, longer hospital stays, slower recovery, and depression, along with pregnancy risks such as preterm birth and low birth weight. Furthermore, infants born to iron-deficient mothers are at risk for delayed childhood growth and cognitive development. Preoperative optimization is crucial for improving clinical outcomes, as iron deficiency anemia accounts for over 80% of anemia cases in these patients.

Traditionally, oral (PO) iron supplementation has been the standard approach recommended by the American College of Obstetrics and Gynecology (ACOG) for preventing and addressing iron deficiency due to its simplicity and cost-effectiveness. However, it is marred by poor adherence to therapy and a high incidence of gastrointestinal side effects. While numerous publications have documented the safety and efficacy of intravenous (IV) iron, its utilization remains limited. Currently, IV iron is primarily reserved for patients who exhibit intolerance or an inadequate response to oral therapy. At our institution, we have taken proactive steps by administering IV iron infusions to many of our patients at an earlier gestational age, given the high rate of non-compliance with oral iron therapy. Our hypothesis proposes that individuals with iron deficiency anemia, defined as a serum ferritin level of less than 30 ng/mL (with 92% sensitivity and 98% specificity compared to hemoglobin (Hgb) levels), who receive IV iron infusions, will achieve higher Hgb levels upon admission and experience reduced rates of blood transfusions.

This study aims to assess the impact of IV iron infusions on pregnant patients with iron deficiency anemia. We hope that implementing this study will help improve overall population health. We hypothesize that individuals with iron deficiency anemia who receive IV iron infusions will attain higher Hgb levels at the time of admission and experience reduced rates of blood transfusions at the time of delivery.

After obtaining the patient's consent, they will be randomized into either of the two treatment options. All odd numbers will be in the oral iron group and even numbers enrolled into the IV iron group. We intend to administer Ferrous sulfate 325 mg orally every other day on an empty stomach with lemon/orange water, as numerous randomized control trials have demonstrated that increasing the iron dose does not lead to improved efficacy. Venofer 200 mg will be given every other day until the patient reaches their calculated iron deficit. The dose of IV iron will be calculated according to the Ganzoni formula: total iron dose (mg) = body weight (kg) x (target Hgb - baseline Hgb (g/dL)) × 0.24 + 500 mg. Our target Hgb will be 11.0 g/dL.

Patients will be given a symptom questionnaire at the time of enrollment to fill out. We will analyze the patient's ferritin, iron, total iron binding capacity (TIBC), Hgb level, mean corpuscular volume (MCV), and Hgb electrophoresis, which are routinely obtained on the first visit with prenatal labs. Four weeks after initiating treatment, patients will fill out a symptom and side effect questionnaire, and if on PO iron, their compliance will be assessed. Complete blood count (CBC) and iron studies will be repeated at that time. Other patient information such as admission CBC, post-delivery CBC, height, weight, body mass index (BMI), age, parity, gestational age at delivery, quantitative blood loss, route of delivery, need for blood transfusion, number of IV iron infusions, fetal birth weight, and antepartum/intrapartum/postpartum complications such as diabetes, preeclampsia/eclampsia, chorioamnionitis, and hemorrhage, etc., neonatal intensive care unit (NICU) admission as well as Edinburgh depression screening results, will be obtained from medical records. This information will be used for secondary outcomes analysis and to ensure there are no confounding factors. Statistical comparisons between groups will be performed using the two-way T-test followed by Tukey's test, or post hoc Student-Newman-Keuls tests. A P < .05 will be considered a statistically significant difference among groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Ferritin level < 30 ng/mL
* Singe gestation
* Gestational age up to 36 weeks as iron therapy after this has shown to be not beneficial at time of delivery. We will still plan to treat patients > 36 weeks but not include them in the final analysis
* Plan to delivery at Arrowhead Regional Medical Center (ARMC)

Exclusion Criteria:

* Maternal age < 18 years of age
* Incarcerated patients
* Multifetal gestation
* Acute liver/kidney disease
* Active infections
* Known hematological malignancy
* Other causes of anemia such as alpha/beta thalassemia, sickle cell disease, Folate/B12 deficiency, and anemia of chronic diseases
* Known hypersensitivity with IV iron
* Severe symptoms of anemia requiring blood transfusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin difference | Hemoglobin level obtained prior to treatment and then 4 weeks later
  Change in hemoglobin level after intervention, larger difference mean more improvement in Hgb
Ferritin difference | Ferritin level obtained prior to treatment and then 4 weeks later
  Change in ferritin level after intervention, larger difference mean more improvement in ferritin level
Delivery Hemoglobin | Obtained at time of delivery
  Comparing pre-delivery hemoglobin levels
Rates of blood transfusion | At time of delivery until 6 weeks postpartum
  Comparing rates of blood transfusion at time of delivery between the 2 groups. The number of units transfused will be collected and compared among the groups
Symptoms | 4 weeks
  Comparing number of anemia symptoms before and after treatment. There are 11 anemia symptoms on the questionnaire. Using a Likert scale from 0 (no symptoms) to 5 (severe symptoms) patient mark each one. The score is totaled up and can range from 0-55.

SECONDARY OUTCOMES:
Preterm delivery | At the time of delivery
  Comparing hemoglobin levels to gestational age at delivery
Depression | Duration of the pregnancy (up to 40 weeks) and up to 2 months postpartum
  Edinburgh postnatal depression scale at first prenatal visit and postpartum. 10 questions with total score between 0-30. Higher score indicated increase risk for depression.
Birthweight | At time of delivery
  Comparing birthweight to hemoglobin levels at time of admission

CONTACTS AND LOCATIONS:
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Froessler B, Palm P, Weber I, Hodyl NA, Singh R, Murphy EM. The Important Role for Intravenous Iron in Perioperative Patient Blood Management in Major Abdominal Surgery: A Randomized Controlled Trial. Ann Surg. 2016 Jul;264(1):41-6. doi: 10.1097/SLA.0000000000001646. PMID 26817624
- [Background] Anemia in Pregnancy: ACOG Practice Bulletin, Number 233. Obstet Gynecol. 2021 Aug 1;138(2):e55-e64. doi: 10.1097/AOG.0000000000004477. PMID 34293770
- [Background] Achebe MM, Gafter-Gvili A. How I treat anemia in pregnancy: iron, cobalamin, and folate. Blood. 2017 Feb 23;129(8):940-949. doi: 10.1182/blood-2016-08-672246. Epub 2016 Dec 29. PMID 28034892
- [Background] Tigga MP, Debbarma AP. A comparative study to evaluate oral iron and intravenous iron sucrose for treatment of anemia in pregnancy in a poor socioeconomic region of Northeast India. Tzu Chi Med J. 2019 Jul 24;32(3):258-261. doi: 10.4103/tcmj.tcmj_99_19. eCollection 2020 Jul-Sep. PMID 32955516
- [Background] Chua S, Gupta S, Curnow J, Gidaszewski B, Khajehei M, Diplock H. Intravenous iron vs blood for acute post-partum anaemia (IIBAPPA): a prospective randomised trial. BMC Pregnancy Childbirth. 2017 Dec 19;17(1):424. doi: 10.1186/s12884-017-1596-x. PMID 29258541
- [Result] Ng O, Keeler BD, Mishra A, Simpson JA, Neal K, Al-Hassi HO, Brookes MJ, Acheson AG. Iron therapy for preoperative anaemia. Cochrane Database Syst Rev. 2019 Dec 7;12(12):CD011588. doi: 10.1002/14651858.CD011588.pub3. PMID 31811820
- [Result] Nicholls G, Mehta R, McVeagh K, Egan M. The Effects of Intravenous Iron Infusion on Preoperative Hemoglobin Concentration in Iron Deficiency Anemia: Retrospective Observational Study. Interact J Med Res. 2022 Feb 3;11(1):e31082. doi: 10.2196/31082. PMID 35113024
- [Result] Lewkowitz AK, Stout MJ, Cooke E, Deoni SC, D'Sa V, Rouse DJ, Carter EB, Tuuli MG. Intravenous versus Oral Iron for Iron-Deficiency Anemia in Pregnancy (IVIDA): A Randomized Controlled Trial. Am J Perinatol. 2022 Jun;39(8):808-815. doi: 10.1055/s-0041-1740003. Epub 2021 Nov 28. PMID 34839481
- [Result] Wong L, Smith S, Gilstrop M, Derman R, Auerbach S, London N, Lenowitz S, Bahrain H, McClintock J, Auerbach M. Safety and efficacy of rapid (1,000 mg in 1 hr) intravenous iron dextran for treatment of maternal iron deficient anemia of pregnancy. Am J Hematol. 2016 Jun;91(6):590-3. doi: 10.1002/ajh.24361. Epub 2016 Apr 13. PMID 26971581
- [Result] Hansen R, Sommer VM, Pinborg A, Krebs L, Thomsen LL, Moos T, Holm C. Intravenous ferric derisomaltose versus oral iron for persistent iron deficient pregnant women: a randomised controlled trial. Arch Gynecol Obstet. 2023 Oct;308(4):1165-1173. doi: 10.1007/s00404-022-06768-x. Epub 2022 Sep 15. PMID 36107229
- [Result] Govindappagari S, Burwick RM. Treatment of Iron Deficiency Anemia in Pregnancy with Intravenous versus Oral Iron: Systematic Review and Meta-Analysis. Am J Perinatol. 2019 Mar;36(4):366-376. doi: 10.1055/s-0038-1668555. Epub 2018 Aug 19. PMID 30121943
- [Result] Stoffel NU, Zeder C, Brittenham GM, Moretti D, Zimmermann MB. Iron absorption from supplements is greater with alternate day than with consecutive day dosing in iron-deficient anemic women. Haematologica. 2020 May;105(5):1232-1239. doi: 10.3324/haematol.2019.220830. Epub 2019 Aug 14. PMID 31413088

DOCUMENTS (1):
  • Informed Consent Form (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT06366698/ICF_000.pdf